CLINICAL TRIAL: NCT02191306
Title: Utilizing Computed Tomographic Angiography to Evaluate Coronary Artery Disease in Patients on Long-Term Antiretroviral Therapy
Status: Completed | Type: Observational
Sponsor: Florida State University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00000446
Record Dates: First submitted 2014-07-14; First posted 2014-07-16 (Estimated); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Evaluate the Relationship Between HIV Medications and Coronary Atherosclerosis
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week

GROUPS / COHORTS (2):
- HIV Positive Patients (Study Group)
- Non HIV Positive Patients (Control)

SUMMARY:
Utilizing Computed Tomographic Angiography to Evaluate Coronary Artery Disease in Patients on Long-Term Antiretroviral Therapy

Intro:

It is well known that HIV treated with antiretroviral drugs increases the risk for coronary artery disease. Studies have documented this with various methods including analyzing the effects of retroviral therapy on cardiac risk factors such as diabetes, lipids and hypertension. Still other studies have looked at carotid and brachial artery intimal thickness. Our study, then, aims to evaluate the relationship between HIV medications and coronary atherosclerosis using a novel method. Coronary artery CT angiography is a relatively new diagnostic procedure to evaluate heart disease in cardiac patients. We will apply this test to HIV patients on longstanding antiretroviral therapy to directly examine their coronary arteries to assess heart disease.

Hypothesis:

We hypothesize that HIV patients on antiretroviral therapy will have increased coronary artery disease compared to the general population.

Methods:

This project will be conducted in collaboration between Florida Heart Center and Associates in infectious Disease - two communities based infectious disease and cardiology practices. We will identify all the HIV positive patients seen within a 1 month timeframe at the infectious disease office. These patients will then be filtered by our exclusion/inclusion criteria. After obtaining informed consent, we will draw blood from each patient to gather lab values such as A1C, cholesterol, inflammatory markers, and other markers associated with coronary artery disease. Each enrolled patient will then schedule and receive a 64 slide coronary CTA at Florida Heart Center. The results of the CTA scans will be categorized in mild, moderate, and severe coronary artery disease. The data, then, will consist of the parameters measured on blood work, and the results of the coronary CTA.

Inclusion Criteria:

1. Patients aged 35 to 50 with HIV and on retroviral therapy for at least 5 years.

Exclusion Criteria:

1. Patients with prior documented coronary artery disease, heart attack, stent placement, or heart surgery.

Statistical Analysis:

We will conduct a multivariate analysis on the cardiac risk factors taken from patient history and the bloodwork (diabetes, lipids etc) to correlate them with the results of the CTA. We will also conduct basic analysis to support our hypothesis that long term antiretroviral therapy increases coronary artery disease.

Funding:

The bloodwork and CTA tests ordered in this study will be payed for by insurance companies where available. In cases where insurance companies will not pay, Florida Heart Center will pay for the CTA tests and Associates in infectious Disease will fund the bloodwork.

Humans Subjects Protection:

This will be a projective chart review study that will require access to protected health information. Thus, we will seek full IRB approval from the FSU IRB committee with informed consent. An informed consent document will be given to each patient explaining all the risks and benefits of the study in addition to the methods. Recruitment will be done by an office staff or medical assistant not on the research team. After patient recruitment, their medical records will be flagged for study and they will undergo the required testing. At completion of testing, their results will be recorded in the final data sheet, and their medical record will no longer be flagged for study. No identifying data will be recorded in the final data sheet, and the data will be stored in an encrypted excel sheet on a secure password protected personal laptop running antivirus and firewall. Third parties (such as family members) will not have access to any research data regardless of authorizations received from the study subjects. All the test results and labwork performed for the study will go into the patient's individual medical record at their respective offices. Thus, if an authorized third party wishes to view any test results, they can do so via the normal methods at the doctor's office.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 35 to 50 with HIV and on retroviral therapy for at least 5 years

Exclusion Criteria:

* Patients with prior documented coronary artery disease, heart attack, stent placement, or heart surgery.

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients aged 35 to 50 with HIV and on antiretroviral therapy for at least 5 years. These patients also cannot have any documented history of coronary artery disease or cardiac interventions.
Sampling Method: Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Calcium Score Measured from CT Angiography | 1 Day
  Each CT Scan was analyzed and a calcium score was associate with each plaque lesion in the coronary arteries. This score correlates with the presence of coronary artery disease in the patient.
Increased Inflammatory Markers in Bloodwork | 1 Day
  The blood work taken from each HIV positive patient was run with a cardiovascular inflammatory marker panel which gave the researchers another measure of coronary artery disease

SECONDARY OUTCOMES:
Increased Inflammatory Markers on Lab Panel | 1 Day
  The blood work taken from each HIV positive patient was run with a cardiovascular inflammatory marker panel which gave the researchers another measure of coronary artery disease

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Associates in Infectious Disease, Ft. Pierce, Florida
  - Florida Heart Center, Ft. Pierce, Florida

REFERENCES:
- [Background] Lo J, Abbara S, Shturman L, Soni A, Wei J, Rocha-Filho JA, Nasir K, Grinspoon SK. Increased prevalence of subclinical coronary atherosclerosis detected by coronary computed tomography angiography in HIV-infected men. AIDS. 2010 Jan 16;24(2):243-53. doi: 10.1097/QAD.0b013e328333ea9e. PMID 19996940
- [Background] Ross AC, Rizk N, O'Riordan MA, Dogra V, El-Bejjani D, Storer N, Harrill D, Tungsiripat M, Adell J, McComsey GA. Relationship between inflammatory markers, endothelial activation markers, and carotid intima-media thickness in HIV-infected patients receiving antiretroviral therapy. Clin Infect Dis. 2009 Oct 1;49(7):1119-27. doi: 10.1086/605578. PMID 19712036
- [Background] Fitch KV, Srinivasa S, Abbara S, Burdo TH, Williams KC, Eneh P, Lo J, Grinspoon SK. Noncalcified coronary atherosclerotic plaque and immune activation in HIV-infected women. J Infect Dis. 2013 Dec 1;208(11):1737-46. doi: 10.1093/infdis/jit508. Epub 2013 Sep 16. PMID 24041790
- See also: Related Info — http://www.hopkinsmedicine.org/news/media/releases/johns_hopkins_study_shows_link_between_hiv_infection_and_coronary_artery_disease
- See also: Related Info — http://www.uptodate.com/contents/cardiac-and-vascular-disease-in-hiv-infected-patients